CLINICAL TRIAL: NCT00584103
Title: Evaluation of an Inexpensive Upper Extremity Prosthesis
Brief Title: Evaluation of Upper Extremity Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORTHDH 07; 13099 (Other: University of Oklahoma Health Sciences Center)
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Transradial Amputation
Keywords: transradial amputation; prosthesis; prefabricated prosthesis; inexpensive; custom prosthesis; adult transradial amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Beta P Experimental (Experimental): Subjects will be fitted with the inexpensive prosthesis model from Prestige Healthcare Technologies. Then the terminal device will be fitted and evaluated using the NYU trans-radial prosthesis checkout form.
  Interventions: Device: Beta P Experimental
- Alpha P Control (Other): Subjects will be fitted with a terminal device with their current prosthesis and evaluated using the NYU trans-radial prosthesis checkout form.
  Interventions: Device: Alpha P Control

INTERVENTIONS:
Device: Alpha P Control — Subjects will be fitted with a terminal device with their current prosthesis and evaluated using the NYU trans-radial prosthesis checkout form.
  Other Names: Standard/Current Prosthesis
  Arms: Alpha P Control
Device: Beta P Experimental — Subjects will be fitted with the inexpensive prosthesis model from Prestige Healthcare Technologies. Then the terminal device will be fitted and evaluated using the NYU trans-radial prosthesis checkout form.
  Other Names: Inexpensive Prosthesis
  Arms: Beta P Experimental

SUMMARY:
The purpose of this study is to evaluate a design of prosthesis that is inexpensive and able to fit a multitude of individuals. This may offer an off the shelf item for those that cannot afford a customized prosthesis, or wish to have an inexpensive spare.

DETAILED DESCRIPTION:
A prospective study will be done on an inexpensive below elbow upper extremity prosthesis. Prestige Healthcare Technologies Ltd. has developed a prosthesis that is easily and inexpensively fabricated. The prosthesis is similar to a fitting frame used by some prosthetists in trial fits to ensure proper length and angulation of the terminal device. The prosthesis consists of two pieces of aluminum bar stock running midline the length of the residual limb. One bar is located anteriorly, the other posteriorly. A terminal device will be placed in the receiver on the distal end of the prosthesis. An aluminum band will connect the anterior and posterior bar stock for structural stability. A finished figure of eight harness will be utilized for control and suspension of the prosthesis. The research performed will be noninvasive. The check out will be based on the New York University (NYU) trans-radial prosthesis checkout form. Prestige Healthcare Technologies has donated an adult size trans-radial prosthesis to be utilized for this study.

Each patient will serve as their own control group. The control group will be considered using the same guidelines for testing function of the patient's current prosthesis, which we will refer to as alpha P. The patient will then be fitted with the inexpensive model, which we will refer to as beta P. The results will be compared to the NYU standard as well as comparing between the results of alpha P and beta P. Beta P will be the same prosthesis personalized for subjects with the harness adjusted to properly fit each individual.

The benefit of this study may provide an inexpensive versatile alternative to the current below elbow prosthesis. This version may be utilized as a spare prosthesis while the patient is unable to use his primary prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with unilateral transradial amputation
* Neurologically intact
* At least 6 months post amputation surgery
* Skin integrity intact without ulceration

Exclusion Criteria:

* Bilateral upper extremity amputees
* Patients that are insensate
* Patients with poor skin integrity
* Patients whose residual limb lengths preclude them from using the transradial prosthesis that is being evaluated

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-01; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
correct application and maintenance of position of device | 1 day -- time it takes to take measurements and make observations

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hunt, B.S., C.O., Principal Investigator — University of Oklahoma Health Sciences Center Department of Orthopedic Surgery & Rehabilitation, Division of Orthotics & Prosthetics
Locations (1):
- University of Oklahoma Health Sciences Center, O'Donoghue Orthotics & Prosthetics Clinic, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No